CLINICAL TRIAL: NCT01139281
Title: The Protective Effect of Ginkgo Biloba Extract on Cisplatin-Induced Ototoxicity in Humans Beings Evaluated by Distortion Product Otoacoustic Emissions
Brief Title: The Protective Effect of Ginkgo Biloba Extract on Cisplatin-induced Ototoxicity in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Mirela Alves Dias, University of Brasilia - Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEPSESDF-024-07
Record Dates: First submitted 2010-06-01; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-05

CONDITIONS: Ototoxicity; Hearing Loss
Keywords: Ear protection; Ginkgo Biloba Extract; Distortion-product otoacoustic emission; Ototoxicity; Cisplatin
MeSH Terms: conditions — Ototoxicity; Hearing Loss | interventions — Ginkgo biloba extract; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): The Study Group(SG) received Ginkgo biloba extract(GBE761)(240mg/day)plus cisplatin(CDDP)
  Interventions: Drug: Ginkgo Biloba Extract (GBE761)
- Control Group(CG) (Placebo Comparator): The Control Group received Placebo plus CDDP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginkgo Biloba Extract (GBE761) — The subjects were randomized and allocated in two groups: Control Group(CG) and Study Group(SG). the study group received GBE761(120mg twice a day) plus cisplatin and was guided to ingest GBE761 just before initial cisplatin dosage. The maximum cumulative cisplatin dosage was 300mg/m². They were followed up for ninety days. Comparisons were made between baseline distortion-product otoacoustic emissions measurements and those DPOAE records after maximum cumulative cisplatin dosage.
  Other Names: Study Group
  Arms: Study Group
Drug: Placebo — The subjects were randomized and allocated in two groups: control group and study group. The control group received placebo plus cisplatin and was guided to ingest Placebo just before initial cisplatin dosage. The maximum cumulative cisplatin dosage was 300mg/m². They were followed up for ninety days. Comparisons were made between baseline distortion-product otoacoustic emissions measurements and those DPOAE records after maximum cumulative cisplatin dosage.
  Other Names: Control Group
  Arms: Control Group(CG)

SUMMARY:
The proposal of this study was to evaluate in human beings, using distortion product otoacoustic emission (DPOAE) test, the action of ginkgo biloba extract (GBE761)as a possible ear protective against cisplatin (CDDP) induced hearing loss.

DETAILED DESCRIPTION:
The ototoxicity is an alteration caused by drugs that compromises the auditory and vestibular functions. The cisplatin (CDDP) is a potent antineoplastic agent used for the treatment of cancer in both adults and children although it has several side effects. Current opinion is that cisplatin ototoxicity occurs due to alterations in the antioxidant system of the outer hair cells (OHC) of the cochlea. The distortion-product otoacoustic emissions (DPOAE) has been showed to be a sensitive test for diagnosis of OHC injury and has been used for monitoring treatment with ototoxic drugs. Because of their antioxidant properties, the ginkgo biloba extract (GBE761) was evaluated in human beings as a possible ear protective against cisplatin induced hearing loss, using DPOAE test.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of eighteen
* Patients that will begin treatment with cisplatin
* No prior treatment with cisplatin

Exclusion Criteria:

* Individuals with middle ear, cochlear or retrocochlear disease
* Presence of changes in pure tone audiometry and/or distortion-product otoacoustic emissions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
the effect of GBE761 as a possible protector against cisplatin (CDDP) induced hearing loss was evaluated through the DPOAE. Comparisons were made between baseline measurements and those records after maximum cumulative CDDP dosage. | the patients were followed about ninety days
  The protective effect of GBE761 on CDDP induced ototoxicity in human beings was evaluated with DPOAE mean amplitudes and signal-to-noise ratio (SNR) values at in the frequencies ranging from 1 to 8KHz in the study and control groups, between before and after cumulative CDDP injections, in order to evaluate the significant differences in DPOAE results, and so to differentiate hearing status ( normal hearing or hearing loss) while the subjects were taking GBE or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Mirela A Dias, Principal Investigator — University of Brasilia; Carlos CP Oliveira, Study Chair — University of Brasilia
Locations (1):
- Hospital de Base do Distrito Federal (HBDF), Brasília, Federal District, Brazil

REFERENCES:
- [Background] Biro K, Noszek L, Prekopp P, Nagyivanyi K, Geczi L, Gaudi I, Bodrogi I. Characteristics and risk factors of cisplatin-induced ototoxicity in testicular cancer patients detected by distortion product otoacoustic emission. Oncology. 2006;70(3):177-84. doi: 10.1159/000093776. Epub 2006 Jun 2. PMID 16757924
- [Background] Blakley BW, Myers SF. Patterns of hearing loss resulting from cis-platinum therapy. Otolaryngol Head Neck Surg. 1993 Sep;109(3 Pt 1):385-91. doi: 10.1177/019459989310900302. PMID 8414553
- [Background] Bridi R, Crossetti FP, Steffen VM, Henriques AT. The antioxidant activity of standardized extract of Ginkgo biloba (EGb 761) in rats. Phytother Res. 2001 Aug;15(5):449-51. doi: 10.1002/ptr.814. PMID 11507743
- [Background] Christen Y, Maixent JM. What is Ginkgo biloba extract EGb 761? An overview--from molecular biology to clinical medicine. Cell Mol Biol (Noisy-le-grand). 2002 Sep;48(6):601-11. PMID 12396070
- [Background] Dhooge I, Dhooge C, Geukens S, De Clerck B, De Vel E, Vinck BM. Distortion product otoacoustic emissions: an objective technique for the screening of hearing loss in children treated with platin derivatives. Int J Audiol. 2006 Jun;45(6):337-43. doi: 10.1080/14992020600582117. PMID 16777780
- [Background] Gardner CD, Zehnder JL, Rigby AJ, Nicholus JR, Farquhar JW. Effect of Ginkgo biloba (EGb 761) and aspirin on platelet aggregation and platelet function analysis among older adults at risk of cardiovascular disease: a randomized clinical trial. Blood Coagul Fibrinolysis. 2007 Dec;18(8):787-93. doi: 10.1097/MBC.0b013e3282f102b1. PMID 17982321
- [Background] Gorga MP, Neely ST, Ohlrich B, Hoover B, Redner J, Peters J. From laboratory to clinic: a large scale study of distortion product otoacoustic emissions in ears with normal hearing and ears with hearing loss. Ear Hear. 1997 Dec;18(6):440-55. doi: 10.1097/00003446-199712000-00003. PMID 9416447
- [Background] Gorga MP, Stover L, Neely ST, Montoya D. The use of cumulative distributions to determine critical values and levels of confidence for clinical distortion product otoacoustic emission measurements. J Acoust Soc Am. 1996 Aug;100(2 Pt 1):968-77. doi: 10.1121/1.416208. PMID 8759950
- [Background] Hatzopoulos S, Di Stefano M, Campbell KC, Falgione D, Ricci D, Rosignoli M, Finesso M, Albertin A, Previati M, Capitani S, Martini A. Cisplatin ototoxicity in the Sprague Dawley rat evaluated by distortion product otoacoustic emissions. Audiology. 2001 Sep-Oct;40(5):253-64. PMID 11688544
- [Background] Hibatallah J, Carduner C, Poelman MC. In-vivo and in-vitro assessment of the free-radical-scavenger activity of Ginkgo flavone glycosides at high concentration. J Pharm Pharmacol. 1999 Dec;51(12):1435-40. doi: 10.1211/0022357991777083. PMID 10678500
- [Background] Huang T, Cheng AG, Stupak H, Liu W, Kim A, Staecker H, Lefebvre PP, Malgrange B, Kopke R, Moonen G, Van De Water TR. Oxidative stress-induced apoptosis of cochlear sensory cells: otoprotective strategies. Int J Dev Neurosci. 2000 Apr-Jun;18(2-3):259-70. doi: 10.1016/s0736-5748(99)00094-5. PMID 10715580
- [Background] Rybak LP, Husain K, Morris C, Whitworth C, Somani S. Effect of protective agents against cisplatin ototoxicity. Am J Otol. 2000 Jul;21(4):513-20. PMID 10912697
- [Background] Kaltenbach JA, Church MW, Blakley BW, McCaslin DL, Burgio DL. Comparison of five agents in protecting the cochlea against the ototoxic effects of cisplatin in the hamster. Otolaryngol Head Neck Surg. 1997 Nov;117(5):493-500. doi: 10.1016/S0194-59989770020-2. PMID 9374173
- [Background] Kobuchi H, Droy-Lefaix MT, Christen Y, Packer L. Ginkgo biloba extract (EGb 761): inhibitory effect on nitric oxide production in the macrophage cell line RAW 264.7. Biochem Pharmacol. 1997 Mar 21;53(6):897-903. doi: 10.1016/s0006-2952(96)00873-8. PMID 9113109
- [Background] Meyerhoff WL, Maale GE, Yellin W, Roland PS. Audiologic threshold monitoring of patients receiving ototoxic drugs. Preliminary report. Ann Otol Rhinol Laryngol. 1989 Dec;98(12 Pt 1):950-4. doi: 10.1177/000348948909801206. PMID 2589763
- [Background] Palomar Garcia V, Abdulghani Martinez F, Bodet Agusti E, Andreu Mencia L, Palomar Asenjo V. Drug-induced otoxicity: current status. Acta Otolaryngol. 2001 Jul;121(5):569-72. doi: 10.1080/00016480121545. PMID 11583387
- [Background] Campbell K. Ototoxicity: understanding oxidative mechanisms. J Am Acad Audiol. 2003 Apr;14(3):121-3. doi: 10.3766/jaaa.14.3.2. No abstract available. PMID 14558530
- [Background] Campbell KC, Durrant J. Audiologic monitoring for ototoxicity. Otolaryngol Clin North Am. 1993 Oct;26(5):903-14. PMID 8233496
- [Background] Diamond BJ, Shiflett SC, Feiwel N, Matheis RJ, Noskin O, Richards JA, Schoenberger NE. Ginkgo biloba extract: mechanisms and clinical indications. Arch Phys Med Rehabil. 2000 May;81(5):668-78. doi: 10.1016/s0003-9993(00)90052-2. PMID 10807109
- [Background] Franklin DJ, McCoy MJ, Martin GK, Lonsbury-Martin BL. Test/retest reliability of distortion-product and transiently evoked otoacoustic emissions. Ear Hear. 1992 Dec;13(6):417-29. doi: 10.1097/00003446-199212000-00008. PMID 1487104
- [Background] Bonfils P, Avan P. Distortion-product otoacoustic emissions. Values for clinical use. Arch Otolaryngol Head Neck Surg. 1992 Oct;118(10):1069-76. doi: 10.1001/archotol.1992.01880100061014. PMID 1389058
- [Background] Kemp DT, Ryan S, Bray P. A guide to the effective use of otoacoustic emissions. Ear Hear. 1990 Apr;11(2):93-105. doi: 10.1097/00003446-199004000-00004. PMID 2340969
- [Background] Kimberley BP. Applications of distortion-product emissions to an otological practice. Laryngoscope. 1999 Dec;109(12):1908-18. doi: 10.1097/00005537-199912000-00003. PMID 10591346
- [Background] Knight KR, Kraemer DF, Winter C, Neuwelt EA. Early changes in auditory function as a result of platinum chemotherapy: use of extended high-frequency audiometry and evoked distortion product otoacoustic emissions. J Clin Oncol. 2007 Apr 1;25(10):1190-5. doi: 10.1200/JCO.2006.07.9723. PMID 17401008
- [Background] Komune S, Asakuma S, Snow JB Jr. Pathophysiology of the ototoxicity of cis-diamminedichloroplatinum. Otolaryngol Head Neck Surg. 1981 Mar-Apr;89(2):275-82. doi: 10.1177/019459988108900226. PMID 6787526
- [Background] Kushner BH, Budnick A, Kramer K, Modak S, Cheung NK. Ototoxicity from high-dose use of platinum compounds in patients with neuroblastoma. Cancer. 2006 Jul 15;107(2):417-22. doi: 10.1002/cncr.22004. PMID 16779793
- [Background] Laurell G, Bagger-Sjoback D. Dose-dependent inner ear changes after i.v. administration of cisplatin. J Otolaryngol. 1991 Jun;20(3):158-67. PMID 1870163
- [Background] Le Bars PL, Kastelan J. Efficacy and safety of a Ginkgo biloba extract. Public Health Nutr. 2000 Dec;3(4A):495-9. doi: 10.1017/s1368980000000574. PMID 11276297
- [Background] Lonsbury-Martin BL, Whitehead ML, Martin GK. Clinical applications of otoacoustic emissions. J Speech Hear Res. 1991 Oct;34(5):964-81. doi: 10.1044/jshr.3405.964. PMID 1749251
- [Background] Mahadevan S, Park Y. Multifaceted therapeutic benefits of Ginkgo biloba L.: chemistry, efficacy, safety, and uses. J Food Sci. 2008 Jan;73(1):R14-9. doi: 10.1111/j.1750-3841.2007.00597.x. PMID 18211362
- [Background] Maitra I, Marcocci L, Droy-Lefaix MT, Packer L. Peroxyl radical scavenging activity of Ginkgo biloba extract EGb 761. Biochem Pharmacol. 1995 May 26;49(11):1649-55. doi: 10.1016/0006-2952(95)00089-i. PMID 7786306
- [Background] Marcocci L, Packer L, Droy-Lefaix MT, Sekaki A, Gardes-Albert M. Antioxidant action of Ginkgo biloba extract EGb 761. Methods Enzymol. 1994;234:462-75. doi: 10.1016/0076-6879(94)34117-6. No abstract available. PMID 7808320
- [Background] McKenna DJ, Jones K, Hughes K. Efficacy, safety, and use of ginkgo biloba in clinical and preclinical applications. Altern Ther Health Med. 2001 Sep-Oct;7(5):70-86, 88-90. PMID 11565403
- [Background] Ohlms LA, Lonsbury-Martin BL, Martin GK. The clinical application of acoustic distortion products. Otolaryngol Head Neck Surg. 1990 Jul;103(1):52-9. doi: 10.1177/019459989010300108. PMID 2117731
- [Background] Ozturan O, Jerger J, Lew H, Lynch GR. Monitoring of cisplatin ototoxicity by distortion-product otoacoustic emissions. Auris Nasus Larynx. 1996;23:147-51. doi: 10.1016/s0385-8146(96)80023-x. PMID 8809338
- [Background] Pincemail J, Dupuis M, Nasr C, Hans P, Haag-Berrurier M, Anton R, Deby C. Superoxide anion scavenging effect and superoxide dismutase activity of Ginkgo biloba extract. Experientia. 1989 Aug 15;45(8):708-12. doi: 10.1007/BF01974564. PMID 2547645
- [Background] Probst R, Hauser R. Distortion product otoacoustic emissions in normal and hearing-impaired ears. Am J Otolaryngol. 1990 Jul-Aug;11(4):236-43. doi: 10.1016/0196-0709(90)90083-8. PMID 2240411
- [Background] Ravi R, Somani SM, Rybak LP. Mechanism of cisplatin ototoxicity: antioxidant system. Pharmacol Toxicol. 1995 Jun;76(6):386-94. doi: 10.1111/j.1600-0773.1995.tb00167.x. PMID 7479581
- [Background] Rademaker-Lakhai JM, Crul M, Zuur L, Baas P, Beijnen JH, Simis YJ, van Zandwijk N, Schellens JH. Relationship between cisplatin administration and the development of ototoxicity. J Clin Oncol. 2006 Feb 20;24(6):918-24. doi: 10.1200/JCO.2006.10.077. PMID 16484702
- [Background] Ress BD, Sridhar KS, Balkany TJ, Waxman GM, Stagner BB, Lonsbury-Martin BL. Effects of cis-platinum chemotherapy on otoacoustic emissions: the development of an objective screening protocol. Third place--Resident Clinical Science Award 1998. Otolaryngol Head Neck Surg. 1999 Dec;121(6):693-701. doi: 10.1053/hn.1999.v121.a101567. PMID 10580222
- [Background] Rybak LP, Kelly T. Ototoxicity: bioprotective mechanisms. Curr Opin Otolaryngol Head Neck Surg. 2003 Oct;11(5):328-33. doi: 10.1097/00020840-200310000-00004. PMID 14502062
- [Background] Rybak LP. Mechanisms of cisplatin ototoxicity and progress in otoprotection. Curr Opin Otolaryngol Head Neck Surg. 2007 Oct;15(5):364-9. doi: 10.1097/MOO.0b013e3282eee452. PMID 17823555
- [Background] Rybak LP, Whitworth CA, Mukherjea D, Ramkumar V. Mechanisms of cisplatin-induced ototoxicity and prevention. Hear Res. 2007 Apr;226(1-2):157-67. doi: 10.1016/j.heares.2006.09.015. Epub 2006 Nov 17. PMID 17113254
- [Background] Rybak LP, Whitworth C, Somani S. Application of antioxidants and other agents to prevent cisplatin ototoxicity. Laryngoscope. 1999 Nov;109(11):1740-4. doi: 10.1097/00005537-199911000-00003. PMID 10569399
- [Background] Rybak LP, Ramkumar V. Ototoxicity. Kidney Int. 2007 Oct;72(8):931-5. doi: 10.1038/sj.ki.5002434. Epub 2007 Jul 25. PMID 17653135
- [Background] Rybak LP, Whitworth CA. Ototoxicity: therapeutic opportunities. Drug Discov Today. 2005 Oct 1;10(19):1313-21. doi: 10.1016/S1359-6446(05)03552-X. PMID 16214676
- [Background] Sie KC, Norton SJ. Changes in otoacoustic emissions and auditory brain stem response after cis-platinum exposure in gerbils. Otolaryngol Head Neck Surg. 1997 Jun;116(6 Pt 1):585-92. doi: 10.1016/S0194-59989770232-8. PMID 9215367
- [Background] Singh B, Kaur P, Gopichand, Singh RD, Ahuja PS. Biology and chemistry of Ginkgo biloba. Fitoterapia. 2008 Sep;79(6):401-18. doi: 10.1016/j.fitote.2008.05.007. Epub 2008 Jun 27. PMID 18639617
- [Background] Stavroulaki P, Apostolopoulos N, Segas J, Tsakanikos M, Adamopoulos G. Evoked otoacoustic emissions--an approach for monitoring cisplatin induced ototoxicity in children. Int J Pediatr Otorhinolaryngol. 2001 May 31;59(1):47-57. doi: 10.1016/s0165-5876(01)00455-4. PMID 11376818
- [Background] Stover L, Gorga MP, Neely ST, Montoya D. Toward optimizing the clinical utility of distortion product otoacoustic emission measurements. J Acoust Soc Am. 1996 Aug;100(2 Pt 1):956-67. doi: 10.1121/1.416207. PMID 8759949
- [Background] Toral-Martinon R, Shkurovich-Bialik P, Collado-Corona MA, Mora-Magana I, Goldgrub-Listopad S, Shkurovich-Zaslavsky M. Distortion product otoacoustic emissions test is useful in children undergoing cisplatin treatment. Arch Med Res. 2003 May-Jun;34(3):205-8. doi: 10.1016/S0188-4409(03)00022-5. PMID 14567400
- [Background] Vermorken JB, Kapteijn TS, Hart AA, Pinedo HM. Ototoxicity of cis-diamminedichloroplatinum (II): influence of dose, schedule and mode of administration. Eur J Cancer Clin Oncol. 1983 Jan;19(1):53-8. doi: 10.1016/0277-5379(83)90398-x. PMID 6682776
- [Background] Zorowka PG, Schmitt HJ, Gutjahr P. Evoked otoacoustic emissions and pure tone threshold audiometry in patients receiving cisplatinum therapy. Int J Pediatr Otorhinolaryngol. 1993 Jan;25(1-3):73-80. doi: 10.1016/0165-5876(93)90011-q. PMID 8436482
- [Background] Sockalingam R, Freeman S, Cherny TL, Sohmer H. Effect of high-dose cisplatin on auditory brainstem responses and otoacoustic emissions in laboratory animals. Am J Otol. 2000 Jul;21(4):521-7. PMID 10912698
- [Result] Fukaya H, Kanno H. [Experimental studies of the protective effect of ginkgo biloba extract (GBE) on cisplatin-induced toxicity in rats]. Nihon Jibiinkoka Gakkai Kaiho. 1999 Jul;102(7):907-17. doi: 10.3950/jibiinkoka.102.907. Japanese. PMID 10459293
- [Result] Huang X, Whitworth CA, Rybak LP. Ginkgo biloba extract (EGb 761) protects against cisplatin-induced ototoxicity in rats. Otol Neurotol. 2007 Sep;28(6):828-33. doi: 10.1097/mao.0b013e3180430163. PMID 17450108